CLINICAL TRIAL: NCT03524157
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Preservative-free Ophthalmic Solution PRO-087 Versus Xyel Ofteno® and Systane Ultra®, on the Ocular Surface of Ophthalmologically and Clinically Healthy Subjects
Brief Title: Safety and Tolerability of PRO-087 Versus Xyel Ofteno® and Systane Ultra®, on the Ocular Surface of Healthy Subjects
Acronym: PRO-087/I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOPH087-0616/I
Record Dates: First submitted 2018-04-25; First posted 2018-05-14 (Actual); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye Syndromes; Lubricant Allergy; Tear Disorder
Keywords: Humylub PF; artificial tears; Ophthalmic lubricant; Chondroitin sulfate; Sodium hyaluronate
MeSH Terms: conditions — Dry Eye Syndromes | interventions — chondroitin sulfate, sodium hyaluronate drug combination; polyethylene glycol 400; xanthan gum; Chondroitin Sulfates

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding It will consist in the elimination of the primary label (commercial) in the case of Xyel Ofteno® and Systane Ultra® and the placement of a label identical to the other interventions. Because the bottle in which Systane Ultra® is packaged differs in the color and shape of the lid used by Xyel Ofteno® and PRO-087, a masking will be carried out on the primary packaging which will be identical for the three interventions.The allocation sequence will be generated by personnel assigned. The research center will receive a set of envelopes which will contain the intervention number individually. The envelopes will be identical on the outside. Each of these envelopes will be shown to the participants for their election by the principal investigator or by a designated member of their team.
  The blinding will correspond to the research subject and the principal investigator. In addition, the statistical analysis will be carried out in a blinded manner for the all analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRO-087 (Experimental): Dosage: 1 drop in both eyes, 4 times a day during the waking period per 10 days Active principles: chondroitin sulfate 0.18%, sodium hyaluronate 0.1% ophthalmic solution made by Laboratorios Sophia, S.A. de C.V., transparent solution, free of visible particles in a sterile multi-dose bottle.
  Interventions: Drug: PRO-087
- Xyel Ofteno (Active Comparator): Dosage: 1 drop in both eyes, 4 times a day during the waking period per 10 days, Active principles: Xanthan gum 0.9 mg, sodium chondroitin sulfate 1.0 ophthalmic solution made by Laboratorios Sophia, S.A. de C.V., transparent solution, free of visible particles in a sterile multi-dose bottle.
  Interventions: Drug: Xyel Ofteno
- Systane ultra (Active Comparator): Dosage: 1 drop in both eyes, 4 times a day during the waking period per 10 days Active principles: Polyethylene glycol 400 0.4%, propyleneglycol 0.3%, Ophthalmic solution, multi-dose dropper bottle, made by Alcon Laboratories, Inc.
  Interventions: Drug: Systane Ultra

INTERVENTIONS:
Drug: PRO-087 — The intervention period consists of a therapy with PRO-087administered 4 times a day in the waking period for 10 days. with a security call to day 13.
  Other Names: chondroitin sulfate + sodium hyaluronate; Humylub PF; humylub preservative-free ophthalmic solution; humylub preservative-free ophthalmic solution PF; humylub preservative-free; humylub PF preservative-free; humylub PF ophthalmic solution
  Arms: PRO-087
Drug: Systane Ultra — The intervention period with active comparator drug consists of a therapy with systane administered 4 times a day in the waking period for 10 days. with a security call to day 13.
  Other Names: Polyethylene glycol 400 0.4%, propyleneglycol 0.3%
  Arms: Systane ultra
Drug: Xyel Ofteno — The intervention period with active comparator drug consists of a therapy with Xyel administered 4 times a day in the waking period for 10 days. with a security call to day 13.
  Other Names: Xanthan gum 0.9 mg, sodium chondroitin sulfate
  Arms: Xyel Ofteno

SUMMARY:
Phase I clinical study, to evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-087 versus Xyel Ofteno® and Systane Ultra®, on the ocular surface of ophthalmological and clinically healthy subjects.

Objective: To evaluate the safety and tolerability of the preservative-free formulation PRO-087 manufactured by Laboratorios Sophia S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis:

The ophthalmic solution PRO-087 presents a profile of safety and tolerability similar to comparators in healthy subjects

Methodology:

Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.

DETAILED DESCRIPTION:
Phase I clinical study, to evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-087 versus Xyel Ofteno® and Systane Ultra®, on the ocular surface of ophthalmological and clinically healthy subjects.

Objective: To evaluate the safety and tolerability of the preservative-free formulation PRO-087 manufactured by Laboratorios Sophia S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis:

The ophthalmic solution PRO-087 presents a profile of safety and tolerability similar to comparators in healthy subjects

Methodology:

Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.

Study period:

3 to 4 months

treatment duration: 10 days

Number of patients:

30 subjects, divided into 3 groups,10 subjects (20 eyes) exposed by group.

Diagnosis and main inclusion criteria:

* Systemically and ophthalmologically healthy subjects
* Signed informed consent.
* Age between 18 to 40 years
* Both genders
* Blood tests complete, blood count (BHC), three element blood chemistry (QS) and liver function tests, within normal parameters
* Visual capacity 20/30 or better

Test product, dose and route of administration:

- PRO-087. Chondroitin sulfate 0.18% / 0.1% sodium hyaluronate, ophthalmic solution preservative free. made by Laboratorios Sophia, S.A. of C.V., Zapopan, Jalisco, Mexico.

Dosage: 1 drop 4 times a day during the waking period, both eyes Route of administration: topical ophthalmic.

Reference product, dose and route of administration:

1. Xyel Ofteno®. Xanthan gum 0.09% / Chondroitin sulfate 0.1% / preservative-free ophthalmic solution. made by Laboratorios Sophia, S.A. of C.V., Zapopan, Jalisco, Mexico.

   Dosage: 1 drop 4 times a day during the waking period, both eyes Route of administration: topical ophthalmic.
2. Systane Ultra®. Polyethylene glycol 400 0.4%, propylene glycol 0.3%. made by Alcon Laboratories, Inc.

Dosage: 1 drop 4 times a day during the waking period, both eyes Route of administration: topical ophthalmic.

Evaluation criteria:

Primary security outcome variables:

* Goblet cells density .
* Presence of adverse events.
* Intraocular pressure.
* Visual ability
* Laboratory tests
* Epithelial defects in cornea and conjunctiva.
* Ophthalmological signs: conjunctival hyperemia, chemosis.

Secondary outcome variables:

* Tear film rupture time
* Life signs: heart rate, respiratory frequency systemic blood pressure.
* Subsequent segment

Primary outcome variables of tolerability:

* Burning
* Foreign body sensation
* Itching
* Eye comfort index

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out through the Kruskal-Wallis test for quantitative variables. The difference between the qualitative variables will be analyzed by means of chi square (Chi2). An alpha ≤ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and ophthalmologically healthy subjects
* Signed informed consent.
* Age between 18 to 40 years.
* Both genders
* Blood tests [complete blood count (BHC), three element blood chemistry (QS) and liver function tests (PFH)] within normal parameters
* Visual capacity 20/30 or better

Exclusion Criteria:

* Subjects with a history of hypersensitivity to any of the components of the research products.
* Subject users of topical ophthalmic medications of any pharmacological group.
* Subject users of medication by any other route of administration.
* Women who are pregnant or breastfeeding.
* Women without a history of hysterectomy, oophorectomy or hysterectomy, who do not ensure a hormonal contraceptive method or intrauterine device during the study period.
* Subjects with participation in clinical research studies 90 days prior to inclusion in the present study.
* Diagnosis of liver disease or triple the normal upper value of any of the following liver enzymes: aspartate transferase (AST), alanine transferase (ALT) or bilirubin.
* Inability to attend or answer the evaluations made in each of the visits.
* Positive smoking (specified as cigarette consumption regardless of quantity and frequency)
* Positive alcoholism (specified as the consumption of alcoholic beverages, regardless of quantity and frequency, during the study intervention period).
* Users of contact lenses.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Private Ophthalmological Office, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Started | 10 | 10 | 10
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 1
Not completed — cytology not readable | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Clinical and ophthalmologically healthy subjects who met the inclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (6.8) | 27.2 (6.1) | 28.1 (5.1) | 27.9 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 5 | 6 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 9 | 29
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 10 | 10 | 9 | 29
Intra Ocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHg] | 13.6 (2.3) | 13.5 (2.4) | 13.9 (1.6) | 13.7 (6.3)
tear film breakup (BUT) [Mean (Standard Deviation); unit: seconds] | 8.2 (2.4) | 8.1 (2.1) | 9.3 (2.2) | 8.5 (2.2)
goblet cells [Mean (Standard Deviation); unit: cells /mm2] | 231.4 (103.9) | 244.2 (118.5) | 254.1 (112.9) | 243.2 (111.8)

OUTCOME MEASURES:

1. Primary Outcome: Goblet Cell Density (GCD)
Description: the cells will be measured per square millimeter, it is a continuous variable taken by means of cytology per impression, the normal value is higher than 500 cells per square millimeter
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Mean (Standard Deviation); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 19 | 20 | 17
cells/mm2 | 282.5 (78.6) | 326.8 (125.9) | 291.5 (135.3)
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferior if there are no differences greater than 20%; p = 0.273, Kruskal-Wallis

2. Secondary Outcome: Presence of Adverse Events (AEs)
Description: the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent.
Time Frame: during the 13 days of evaluation, including the safety call (day 13).
Measure: Number; unit: adverse events
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 10
adverse events | 13 | 8 | 7
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p = 0.788, Kruskal-Wallis

3. Secondary Outcome: Intraocular Pressure (IOP)
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
mmHg | 12.80 (1.7) | 12.55 (2.3) | 12.72 (1.5)

4. Secondary Outcome: Epithelial Defects (ED)
Description: The epithelial defects will be evaluated by means of two stains, green lysine and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
eyes
  grade 0 | 19 | 16 | 17
  grade I | 1 | 3 | 1
  grade II | 0 | 1 | 0
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p > 0.05, Chi-squared, Corrected

5. Secondary Outcome: Breakup Time (BUT)
Description: breakup time lacrimal film is a continuous variable that will be measured in seconds, evaluating the time it takes to break it, is done by direct counting and the normality range and mayor to 10 seconds.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
seconds | 8.8 (2.1) | 7.3 (2.1) | 9.6 (2.1)
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p = 0.008, Kruskal-Wallis

6. Secondary Outcome: Conjunctival Hyperemia (CH)
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very mild / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 8
Number analyzed (eyes) | 20 | 20 | 18
cases
  Normal | 19 | 16 | 17
  Very mild | 1 | 3 | 1
  Mild | 0 | 1 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p > 0.05, Chi-squared, Corrected

7. Secondary Outcome: Chemosis
Description: The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
cases | 0 | 0 | 0

8. Secondary Outcome: Ocular Burning (OB)
Description: ocular burning is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale: Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
cases | 4 | 4 | 0
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p > 0.05, Chi-squared, Corrected

9. Secondary Outcome: Foreign Body Sensation (FBS)
Description: Foreign body sensation is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
  Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
cases
  Absent | 20 | 16 | 16
  Very mild | 0 | 4 | 2
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p > 0.05, Chi-squared, Corrected

10. Secondary Outcome: Ocular Pruritus (P)
Description: Ocular pruritus is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
  Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 10)
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (eyes) | 20 | 20 | 18
cases
  Absent | 18 | 16 | 16
  Very mild | 2 | 4 | 2
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRO-087 vs Xyel Ofteno vs Systane Ultra; Test type: Non-Inferiority — it will be considered non-inferiority if there are no differences greater than 20%; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: The monitoring of the adverse events was made throughout the 10 days of intervention of the product and 3 days later by means of a safety telephone call, totaling 13 days of pharmacovigilance.
Description: the treatment is a topical drug, the subjects of investigation with this intervention are not in danger of death.
Arm/Group | PRO-087 | Xyel Ofteno | Systane Ultra
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 4/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-087 (N=10) | Xyel Ofteno (N=10) | Systane Ultra (N=10)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
hypertransaminasemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
ocular burning (Eye disorders) | 4 (4) | 3 (3) | 1 (1)
ocular itching (Eye disorders) | 4 (4) | 2 (2) | 1 (1)
ocular discharge (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
ocular foreign body sensation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
only the sponsor can publish the information held by the research centers, if the principal investigator of a center wishes to publish the information, it must have the written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03524157/Prot_SAP_000.pdf